CLINICAL TRIAL: NCT00737360
Title: Phase II Study of TAS-106 in Patients With Recurrent or Metastatic Head and Neck Cancer Refractory to Platinum Based Chemotherapy
Brief Title: Phase II Study of TAS-106 to Treat Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS106-9905
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — 1-(3-C-ethynylribopentofuranosyl)cytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: TAS-106

INTERVENTIONS:
Drug: TAS-106 — 6.5 mg/m2, IV on day 1 of each 21 day cycle. Number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to determine whether TAS-106 is effective to patients with recurrent or metastatic head and neck cancer refractory to platinum based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ≤ years old at study entry
* Histologically confirmed head and neck carcinoma
* Received prior platinum based regimen and developed disease progression or recurrence
* Measurable disease according to RECIST guidelines

Exclusion Criteria:

* Radiological or clinical evidence of brain involvement or leptomeningeal disease
* ≥ grade 2 peripheral neuropathy
* History of another malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Orleans Street, Baltimore, Maryland
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, Hksar, Hong Kong
- National University Hospital, Lower Kent Ridge Road, Singapore
- National Taiwan University Hospital Department of Oncology, No. 1, Chang-De Street , Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patient enrollment was started from 24/Sep/2008 and terminated as of 30/Sep/2010. In the nasopharyngeal carcinoma (NPC) subgroup and squamous cell carcinoma (SCCHN) subgroup of stage 1, 13 and 14 patients were enrolled, respectively. For both subgroups subsequent enrollment was not reopened for the second stage, thus 27 patients were enrolled.
Period: Overall Study
Arm/Group | TAS-106
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAS-106
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 12
  Taiwan | 1
  Hong Kong | 9
  Singapore | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival(PFS)
Description: PFS was calculated as days from the date of registration until the earliest date of documented disease progression, death, or censoring event.
Time Frame: From the date of registration until the earliest date of documented disease progression, death, or censoring event.
Population: One patient enrolled was discontinued without any post-baseline tumor assessment, therefore, 26 patients were included in the efficacy analyzes.
Measure: Median (95% Confidence Interval); unit: day
Arm/Group | TAS-106
Number analyzed (Participants) | 26
day | 51 [43.0 to 83.0]

2. Secondary Outcome: Antitumor Activity
Description: Antitumor activity was evaluated by measuring the rate of objective response using the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Per RECIST Criteria (V1.0) and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)= CR + PR.", or similar text that was as accurate and appropriate.
Time Frame: Obtain a contrast-enhanced CT scan of the chest, abdomen and pelvis (if clinically indicated) within 28 days prior to study entry and repeat at the end of every 2 courses thereafter.
Population: Antitumor activity was the rate of best overall objective responses(complete response + partial response).
Measure: Number; unit: participants
Arm/Group | TAS-106
Number analyzed (Participants) | 26
participants | 0

3. Secondary Outcome: Overall Survival
Description: Patient survival for both subgroups was followed up every 2 months until 28 Feb 2011.
Time Frame: 12 months after enrollment of the last patient
Measure: Median (95% Confidence Interval); unit: day
Arm/Group | TAS-106
Number analyzed (Participants) | 26
day | 213 [136.0 to 280.0]

4. Secondary Outcome: Safety
Description: Toxicities were evaluated at each course of therapy using the CTCAE ver. 3.0 or a non-CTC grading scale for toxicities that were not covered by the NCI CTC.
Time Frame: Monitor patients for untoward medical events from the time of signed informed consent form, including toxicities from previous treatment and any ongoing or newly reported AEs or SAEs during the 30 days after the last dose of study medication.
Population: All patients who received at least 1 dose of TAS-106 were the primary population for the safety evaluation.
Measure: Number; unit: number of participants
Arm/Group | TAS-106
Number analyzed (Participants) | 27
number of participants | 27

ADVERSE EVENTS:
Time Frame: Adverse events were summarized for all courses of study medication.
Arm/Group | TAS-106
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-106 (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Lymph node abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 1
Hemoglobin decreased (Investigations) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAS-106 (N=27)
Anaemia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 7
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Salivary hypersecretion (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 3
Face oedema (General disorders) | 2
Fatigue (General disorders) | 11
Infusion site discolouration (General disorders) | 2
Injection site reaction (General disorders) | 7
Mucosal inflammation (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Oral candidiasis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 2
Haemoglobin decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 8
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less